CLINICAL TRIAL: NCT01493999
Title: Prasugrel Versus Adjusted High-dose Clopidogrel to TREAT High On-clopidogrel Platelet Reactivity in Acute Coronary Syndrome Patients After PCI
Brief Title: Prasugrel Versus Clopidogrel to TREAT High Platelet Reactivity
Acronym: TREAT-HPR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Daniel Aradi MD, Assisstant Professor, University of Pecs
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PECS-002
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Acute Coronary Syndrome
Keywords: Clopidogrel; prasugrel; HPR; loading dose; maintenance dose; stent thrombosis; platelet reactivity; Coronary intervention; stent implantation
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel arm (Active Comparator): A loading dose of 60 mg prasugrel in patients with HPR after 600 mg clopidogrel.
  Interventions: Drug: Prasugrel
- Clopidogrel reloading (Active Comparator): A maximum of three adjusted loading doses of 600 mg clopidogrel until normal platelet reactivity is achieved in patients with HPR after the first 600 mg clopidogrel.
  Interventions: Drug: Clopidogrel reloading

INTERVENTIONS:
Drug: Clopidogrel reloading — Up to three times 600 mg clopidogrel
  Other Names: Clopidogrel = KARDOGREL
  Arms: Clopidogrel reloading
Drug: Prasugrel — 60 mg prasugrel in patients with HPR
  Other Names: Prasugrel = EFIENT
  Arms: Prasugrel arm

SUMMARY:
MAIN AIM: To compare the pharmacological potency of administering adjusted 600 mg clopidogrel loading doses and 60 mg prasugrel in patients with high on-clopidogrel platelet reactivity (HPR) after PCI.

SECONDARY OBJECTIVES: To define the optimal maintenance dose with both prasugrel (5 mg vs. 10 mg) and clopidogrel (75 mg vs. 150 mg) in patients with HPR for chronic therapy.

DESIGN: Prospective, Randomized, Open-label, Single-center trial.

PRIMARY ENDPOINT: Platelet reactivity measured with Multiplate between clopidogrel and prasugrel arm at day 4.

DETAILED DESCRIPTION:
Study rationale:

After coronary stent implantation, aspirin plus thienopyridine therapy has been proven to be superior to aspirin alone or aspirin plus warfarin in reducing adverse thrombotic events. Due to the lower rate of haematopoietic side effects, once daily administration and faster onset of action, clopidogrel has replaced ticlopidine as the thienopyridine of choice in patients after acute coronary syndrome (ACS) and percutaneous coronary intervention (PCI). However, clopidogrel has many known limitations that might carry important clinical consequences. First, the onset of action of clopidogrel is relatively slow; even a loading dose of 600 mg requires 4-6 hours to achieve the full antiplatelet effect. Second, the antiplatelet potency of clopidogrel is moderate, and platelet reactivity after clopidogrel treatment shows wide inter-patient variability. As a result, a substantial proportion (25-30%) of patients is not receiving proper ADP-receptor inhibition after a fixed-dose clopidogrel regimen and high on-clopidogrel platelet reactivity (HPR) might persist despite clopidogrel administration. In a meta-analysis comprising 20 studies and more than 9,100 patients, those with HPR had a 3.4-fold risk for cardiovascular death, 3-fold risk for myocardial infarction (MI), and 4-fold risk for definite/probable stent thrombosis. According to our current knowledge, the development of HPR is multifactorial: clinical conditions (diabetes, acute coronary syndrome, renal insufficiency, low ejection fraction), laboratory parameters (platelet count, baseline platelet reactivity), patient compliance and genetic predisposition might contribute to the evolution of HPR. (13) Out of these factors, the clinical importance of genetic interaction in clopidogrel-treated subjects was recently emphasized by multiple studies and by a black-boxed warning of the FDA. (14) Based on these, not all clopidogrel-treated patients get the full clinical benefit from clopidogrel therapy and those carrying a loss-of-function allele (LOF: *2 and *3) in the CYP2C19 gene have higher risk to adverse thrombotic events. All these evidences highlight that the currently recommended, fixed-dose clopidogrel treatment is insufficient to prevent the development of HPR and thrombotic events in a significant proportion of patients after PCI.

Up to now, there is limited information on the optimal strategy to overcome HPR. Increasing the maintenance dose of clopidogrel to 150 mg might decrease to rate of HPR; however, it might help in less than 50% of the patients. In one study, the administration of repeated loading doses of 600 mg clopidogrel - based on the results of the vasodilator stimulated phosphoprotein phosphorylation (VASP) assessment - was successful to overcome HPR in 86% of the patients. Importantly, this was the first and only strategy with clopidogrel that was associated with an improvement in the clinical outcome among patients with non-ST segment elevation MI, as the reloaded group had significantly lower rate of major adverse cardiac events compared to conventional fixed dose clopidogrel.

Beyond clopidogrel, there are newer antiplatelet agents that might also be attractive candidates to overcome HPR. Prasugrel is a novel, third-generation thienopyridine that can eliminate many drawbacks of clopidogrel. Compared to clopidogrel, prasugrel leads to a more rapid and greater formation of its active metabolite after absorption as it is not inactivated by the non-specific estherases in the portal circulation. These features result in a more rapid, more uniform and more potent platelet inhibition both after the loading dose and during the maintenance phase with prasugrel compared to even a high-dose of clopidogrel.

However, there is no direct comparison in platelet inhibition between a strategy of administering repeated loading doses of clopidogrel and prasugrel in patients with HPR. Moreover, the optimal maintenance doses of clopidogrel and prasugrel to maintain proper platelet inhibition during the chronic phase of antiplatelet therapy is also unknown.

Thereby, we aim to compare the achievable platelet inhibition after 60 mg prasugrel with adjusted loading doses of 600 mg clopidogrel tailored according to a platelet function assessment in patients after PCI. Moreover, we aim to compare the antiplatelet potency of different clopidogrel (75 vs. 150 mg) and prasugrel (5 mg vs. 10 mg) maintenance doses during the chronic phase of PCI.

Previous work:

Our research team in the University of Pécs, Hungary has been involved in platelet function experiments since more than five years. We described the large inter-individual variability in response to clopidogrel and demonstrated that high on-treatment ADP reactivity is associated with recurrent ischemic events after PCI. We performed a meta-analysis to summarize the clinical significance of high platelet reactivity and described that these patients have 3-fold risk to MI, 4-fold risk to stent thrombosis and 3,4-fold risk for CV death. We also tried to determine the efficacy of 150 mg clopidogrel among patients with high platelet reactivity, together with the clinical and laboratory predictors of good response to the higher maintenance dose. We compared more sophisticated methods of platelet aggregation to light transmission aggregometry.

Study hypothesis:

We hypothesise that prasugrel will provide more rapid and more potent platelet aggregation inhibition compared to repeated loading doses of clopidogrel in patients with HPR after PCI. We also test the efficacy of 5 mg and 10 mg prasugrel as well as 75 and 150 mg clopidogrel in sustaining platelet inhibition in the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-74 years
* PCI with stent implantation due to stable angina or acute coronary syndrome
* Platelet function assessment available 6-24 hours after PCI
* Multiplate-derived ADP-reactivity > 47 U

Exclusion Criteria:

* Age ≥75 years
* Prior TIA or stroke
* Body weight less than 60 kg
* Contraindication for aspirin / thienopyridines
* Severe liver failure (Child Pugh C)
* Need for oral anticoagulation in the following one month
* Planned discontinuation of antiplatelet treatment in one month
* Current bleeding disorder, active bleeding event (Weber positivity)
* Haemoglobin level at presentation < 90 g/l
* Refused informed consent

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
ADP-reactivity between clopidogrel reloading and prasugrel arm | 4 days after randomization
  Multiplate-assessed ADP-reactivity (area under curve, U)

SECONDARY OUTCOMES:
The proportion of patients with HPR | 4 days after randomization
  Multiplate-assessed HPR > 47 U.
ADP-reactivity between clopidogrel and prasugrel arms | 30 days after randomization
  Multiplate-assessed ADP-reactivity (are under curve, U)
The proportion of patients with HPR between clopidogrel and prasugrel arms | 30 days after randomization
  Multiplate-assessed HPR >47 U.
VASP-PRI between clopidogrel and prasugrel patients | 30 days after randomization
  Vasodilator stimulated phosphoprotein phosphorylation assessed with flow cytometer
Cardiovascular death, myocardial infarction or definite/probable stent thrombosis | 30 days after randomization
TIMI major bleeding | 30 days after randomization
  Thrombolysis in Myocardial Infarction-defined major bleeding complications

CONTACTS AND LOCATIONS:
Overall Officials: Dániel Aradi, MD PhD, Principal Investigator — University of Pécs, Heart Institute, Hungary; András Komócsi, MD PhD, Study Director — University of Pécs, Heart Institute, Hungary
Locations (1):
- University of Pécs, Heart Institute, Pécs, Hungary